CLINICAL TRIAL: NCT05583539
Title: A Pilot Study of Thromboelastography Guided Blood Product Transfusion for Patient With Cirrhosis and Upper Gastrointestinal Bleeding
Brief Title: Thromboelastography Guided Blood Product Transfusion for Upper Gastrointestinal Bleeding in Cirrhosis
Acronym: STRATEGIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never IRB approved
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Todd Rice, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 221098
Record Dates: First submitted 2022-10-08; First posted 2022-10-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cirrhosis, Liver; Coagulopathy; GastroIntestinal Bleeding
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders; Gastrointestinal Hemorrhage | interventions — Thrombelastography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Usual Care (No Intervention): Patients will receive usual care at the discretion of their providers.
- Thromboelastography guided resuscitation (Experimental): Patients will undergo thromboelastography testing that will be used by primary providers to guide blood product resuscitation.
  Interventions: Diagnostic Test: Thromboelastography

INTERVENTIONS:
Diagnostic Test: Thromboelastography — Thromboelastography is a viscoelastic test that measures the dynamics of blood clotting on whole blood samples.
  Arms: Thromboelastography guided resuscitation

SUMMARY:
The goal of this clinical trial is to compare resuscitation strategies in patients with cirrhosis and gastrointestinal bleeding. The main question it aims to answer is whether thromboelastography guided resuscitation decreased the amount of fresh frozen plasma patients receive. Patients will receive blood products guided by thromboelastography in the intervention group. Researchers will compare the patients who undergo thromboelastography guided resuscitation to those who receive usual care to see which strategy leads to the use of less blood products, specifically less fresh frozen plasma.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Octreotide order placed for the indication of upper gastrointestinal bleeding in cirrhosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Volume of fresh frozen plasma transfused | From time of randomization to hospital discharge, up to 3 months
  The total volume of fresh frozen plasma transfused

SECONDARY OUTCOMES:
Patients requiring fresh frozen plasma transfusion | From time of randomization to hospital discharge, up to 3 months
  Percentage of patients requiring a fresh frozen plasma transfusion
Volume of platelets and cryoprecipitate transfused | From time of randomization to hospital discharge, up to 3 months
  The total combined volume of platelets and cryoprecipitate transfused
Control of bleeding at 5 days | Measured at 5 days from the time of octreotide order placement
  Percentage of patients who have bleeding controlled at 5 days
Rebleeding at 42 days | The earlier of 42 days from the time of octreotide placement or hospital discharge
  Percentage of patients who experienced in-hospital rebleeding within 42 days
Mortality rate during index hospitalization | From time of randomization to hospital discharge, up to 3 months
  Percentage of patients who died during the index hospitalization

OTHER OUTCOMES:
Rate of transfusion reactions | From time of randomization to hospital discharge, up to 3 months
  Percentage of patients who experienced a transfusion reaction

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rice, MD, Principal Investigator — Vanderbilt University Medical Center

REFERENCES:
- [Background] Lautt WW, Greenway CV. Conceptual review of the hepatic vascular bed. Hepatology. 1987 Sep-Oct;7(5):952-63. doi: 10.1002/hep.1840070527. No abstract available. PMID 3308669
- [Background] D'Amico G, De Franchis R; Cooperative Study Group. Upper digestive bleeding in cirrhosis. Post-therapeutic outcome and prognostic indicators. Hepatology. 2003 Sep;38(3):599-612. doi: 10.1053/jhep.2003.50385. PMID 12939586
- [Background] Tripodi A, Mannucci PM. The coagulopathy of chronic liver disease. N Engl J Med. 2011 Jul 14;365(2):147-56. doi: 10.1056/NEJMra1011170. No abstract available. PMID 21751907
- [Background] Tripodi A, Caldwell SH, Hoffman M, Trotter JF, Sanyal AJ. Review article: the prothrombin time test as a measure of bleeding risk and prognosis in liver disease. Aliment Pharmacol Ther. 2007 Jul 15;26(2):141-8. doi: 10.1111/j.1365-2036.2007.03369.x. PMID 17593061
- [Background] Nanchal R, Subramanian R, Karvellas CJ, Hollenberg SM, Peppard WJ, Singbartl K, Truwit J, Al-Khafaji AH, Killian AJ, Alquraini M, Alshammari K, Alshamsi F, Belley-Cote E, Cartin-Ceba R, Dionne JC, Galusca DM, Huang DT, Hyzy RC, Junek M, Kandiah P, Kumar G, Morgan RL, Morris PE, Olson JC, Sieracki R, Steadman R, Taylor B, Alhazzani W. Guidelines for the Management of Adult Acute and Acute-on-Chronic Liver Failure in the ICU: Cardiovascular, Endocrine, Hematologic, Pulmonary, and Renal Considerations. Crit Care Med. 2020 Mar;48(3):e173-e191. doi: 10.1097/CCM.0000000000004192. PMID 32058387
- [Background] O'Leary JG, Greenberg CS, Patton HM, Caldwell SH. AGA Clinical Practice Update: Coagulation in Cirrhosis. Gastroenterology. 2019 Jul;157(1):34-43.e1. doi: 10.1053/j.gastro.2019.03.070. Epub 2019 Apr 12. PMID 30986390
- [Background] Rout G, Shalimar, Gunjan D, Mahapatra SJ, Kedia S, Garg PK, Nayak B. Thromboelastography-guided Blood Product Transfusion in Cirrhosis Patients With Variceal Bleeding: A Randomized Controlled Trial. J Clin Gastroenterol. 2020 Mar;54(3):255-262. doi: 10.1097/MCG.0000000000001214. PMID 31008867
- [Background] Kumar M, Ahmad J, Maiwall R, Choudhury A, Bajpai M, Mitra LG, Saluja V, Mohan Agarwal P, Bihari C, Shasthry SM, Jindal A, Bhardwaj A, Kumar G, Sarin SK. Thromboelastography-Guided Blood Component Use in Patients With Cirrhosis With Nonvariceal Bleeding: A Randomized Controlled Trial. Hepatology. 2020 Jan;71(1):235-246. doi: 10.1002/hep.30794. Epub 2019 Aug 27. PMID 31148204